CLINICAL TRIAL: NCT01941719
Title: Enhancing Diabetic Foot Education by Viewing Personal Plantar Pressures
Acronym: DFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11447; K23DK081021 (NIH)
Record Dates: First submitted 2013-04-04; First posted 2013-09-13 (Estimated); Results first posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Diabetes Mellitus; Diabetic Neuropathies; Foot Complications
Keywords: Diabetes Mellitus; Diabetic Foot; Diabetic Peripheral Neuropathy; Diabetic Foot Education
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies; Diabetic Foot

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- enhanced foot care education (Experimental): In addition to the standard diabetic foot self-care instruction, the importance of daily foot self-care was reinforced at baseline by viewing personal barefoot plantar pressure in gait
  Interventions: Behavioral: Enhanced foot care education
- Standard Foot Care Education (Active Comparator): Reviewed the standard diabetic foot self-care instructions, including daily foot inspection and proper footwear at all times.
  Interventions: Behavioral: Standard Foot Care Education

INTERVENTIONS:
Behavioral: Enhanced foot care education — In addition to the standard foot care education, personalized, computer-animated plantar pressure maps in both barefoot and in-shoe conditions were demonstrated once at baseline visit. The demonstration includes diabetic foot education on the topic of diabetic neuropathy and how barefoot walking can lead to skin breakdown and ulcer formation, which can lead to infection and eventual amputation. The education also highlights the high plantar pressures experienced by individuals while barefoot versus in-shoe and how proper footwear is necessary in conjunction with other standard self-foot care measures to prevent injury and complications.
  Arms: enhanced foot care education
Behavioral: Standard Foot Care Education — At baseline, a trained staff individually reviewed and dispensed the following brochures: "Prevent diabetes problems: Keep your diabetes under control" (NIH Publication No. 07-4349) and "Prevent diabetes problems: Keep your feet and skin healthy" (NIH Publication No. 07-4282) along with a 1-page summary of each brochure. Also, a 1-page supplementary diabetic shoe wear educational material was reviewed and dispensed. "Keep your diabetes under control" stresses "sugar, blood pressure, and medication control, and nutrition and physical activity, and checking feet daily for cuts, blisters, sores, swelling, redness, or sore toenails." "Keep your skin and feet healthy" emphasizes the importance of checking feet daily, highlighting diabetic foot complications that can arise from neuropathy, poor circulation and dry skin, and the importance of supportive, protective, and accommodative shoewear and annual foot exams.
  Arms: Standard Foot Care Education

SUMMARY:
The purpose of this study is to examine the effectiveness of a novel patient education strategy, compared to a standard diabetic foot education. The proposed diabetic foot care education uses personal computer-animated plantar pressure data to educate patients on why and how they should care for their feet.

DETAILED DESCRIPTION:
Using block randomization, subjects with diabetes were assigned to either the standard or the enhanced education group. The effectiveness of enhanced education was evaluated as measured by foot care behavior score, patient's interpretation of neuropathy scores, and the incidence of diabetic foot complications over a course of 1-year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 21 and 75 years (inclusive)
* Documented type 1 or type 2 diabetes mellitus
* Demonstrates peripheral neuropathy (defined as vibration perception threshold (VPT) ≥ 25 volts at the hallux, as quantified by a BioThesiometer, or unable to perceive a 10 gram Semmes-Weinstein monofilament in one four sites on the feet)
* Able to walk independently without the use of walking aids (cane, crutches, or walker)
* Able to speak and understand English
* Able to understand the information in the informed consent form and willing and able to sign the consent form

Exclusion Criteria:

* Amputation of either foot proximal to midfoot
* Presence of cutaneous ulceration in the lower extremity
* History of or active Charcot neuroarthropathy of either foot
* Severe peripheral vascular disease (ie. ischemic rest pain, 2-block claudication or gangrene)
* End stage kidney disease requiring hemodialysis, stroke, or widespread malignant disease
* Pregnant or nursing
* Life expectancy < 12 months
* Not willing or able to make the required follow-up visits
* Insufficient (corrected) vision to complete the questionnaires

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-05-02 (Actual); Primary Completion 2011-09-07 (Actual); Study Completion 2012-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinsup Song, DPM, PhD, Principal Investigator — Temple University
Locations (1):
- Gait Study Center; Temple University School of Podiatric Medicine, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Foot Care Education: Standard Foot Care Education: At baseline, a trained staff individually reviewed and dispensed the following brochures: "Prevent diabetes problems: Keep your diabetes under control" (NIH Publication No. 07-4349) and "Prevent diabetes problems: Keep your feet and skin healthy" (NIH Publication No. 07-4282). In addition, a 1-page diabetic footwear selection criteria is provided.
- Enhanced Foot Care Education: In addition to the standard diabetic foot educational brochure, the importance of daily foot self-care was reinforced by viewing personal barefoot plantar pressure
Period: Overall Study
Arm/Group | Standard Foot Care Education | Enhanced Foot Care Education
Started | 48 | 51
Month 1 | 43 | 48
Month 3 | 38 | 44
Month 6 | 34 | 42
Month 9 | 29 | 37
Month 12 | 28 | 32
Completed | 28 | 32
Not Completed | 20 | 19
Not completed — Lost to Follow-up | 20 | 19

BASELINE CHARACTERISTICS:
Groups:
- Standard Foot Care Education: Standard Foot Care Education: At baseline, a trained staff individually reviewed and dispensed the following brochures: "Prevent diabetes problems: Keep your diabetes under control" (NIH Publication No. 07-4349) and "Prevent diabetes problems: Keep your feet and skin healthy" (NIH Publication No. 07-4282) along with a 1-page summary of each brochure. Also, a 1-page supplementary diabetic shoe wear educational material was reviewed. "Keep your diabetes under control" stresses "sugar, blood pressure, and medication control, and nutrition and physical activity, and checking feet daily for cuts, blisters, sores, swelling, redness, or sore toenails." "Keep your skin and feet healthy" emphasizes the importance of checking feet daily, highlighting diabetic foot complications that can arise from neuropathy, poor circulation and dry skin, and the importance of supportive, protective, and accommodative shoewear and annual foot exams.
- Enhanced Foot Care Education: In addition to the standard diabetic foot educational brochure, the importance of daily foot self-care was reinforced by viewing personal barefoot plantar pressure
  Personalized, computer-animated plantar pressure maps in both barefoot and in-shoe conditions were demonstrated at baseline visit. Investigator explained how excessive barefoot pressure can lead to skin breakdown and ulcer formation. The education also highlights the benefit of proper footwear and self-foot care measures to prevent injury and complications.
- Total: Total of all reporting groups
Arm/Group | Standard Foot Care Education | Enhanced Foot Care Education | Total
Number analyzed (Participants) | 48 | 51 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (9.5) | 55.9 (10.2) | 54.5 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 30 | 31 | 61
Region of Enrollment [Number; unit: participants]
  United States | 48 | 51 | 99

OUTCOME MEASURES:

1. Primary Outcome: Foot Care Behavior Score
Description: Daily foot inspection - number (& % of participants) of participants who inspect their feet at least daily
Time Frame: baseline, 1, 3,6,9 and 12 months
Population: Fewer participants at follow up visits due to drop out
Measure: Count of Participants; unit: Participants
Groups:
- Standard Foot Care Education: Standard Foot Care Education: At baseline, a trained staff individually reviewed and dispensed the following brochures: "Prevent diabetes problems: Keep your diabetes under control" (NIH Publication No. 07-4349) and "Prevent diabetes problems: Keep your feet and skin healthy" (NIH Publication No. 07-4282). Also, a 1-page supplementary diabetic footwear educational material was reviewed. The aims of education are to emphasize the importance of checking feet daily, highlighting diabetic foot complications that can arise from repetitive trauma and inappropriate footwear in the absence of protective sensation.
Arm/Group | Standard Foot Care Education | Enhanced Foot Care Education
Number analyzed (Participants) | 48 | 51
Participants
  daily foot inspection_baseline | 29 | 36
  daily foot inspection_baselinescore_month 1: number analyzed (Participants) | 43 | 48
  daily foot inspection_baselinescore_month 1 | 33 | 42
  daily foot inspection_baselinescore_month 3: number analyzed (Participants) | 38 | 44
  daily foot inspection_baselinescore_month 3 | 27 | 40
  daily foot inspection_baselinescore_month 6: number analyzed (Participants) | 34 | 42
  daily foot inspection_baselinescore_month 6 | 24 | 35
  daily foot inspection_baselinescore_month 9: number analyzed (Participants) | 29 | 37
  daily foot inspection_baselinescore_month 9 | 19 | 31
  daily foot inspection_baselinescore_month 12: number analyzed (Participants) | 18 | 22
  daily foot inspection_baselinescore_month 12 | 14 | 19
Statistical Analysis 1: Comparison: Standard Foot Care Education vs Enhanced Foot Care Education; A mixed-effect model with repeated measures is used to compare the difference of group over time; Test type: Equivalence — This trial aims to show the enhanced education is no better and no worse than the standard education; p = 0.0770, ANCOVA — significance level set at 0.05; At each follow-up point, multivariate ANCOVA models were used to test for significant changes from the baseline; Mean Difference (Final Values) = -0.1212

2. Primary Outcome: Patient Interpretation of Neuropathy (PIN) Questionnaire
Description: Participants who demonstrated an accurate interpretation of diabetic peripheral neuropathy (id2). The score range from 1 (correct interpretation) to 5 (misinterpretation)
Time Frame: Baseline, months 1, 3, 6, and 12.
Population: Fewer participants in follow up visits due to drop out
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Foot Care Education | Enhanced Foot Care Education
Number analyzed (Participants) | 48 | 51
score on a scale
  id2, baseline | 3.86 (0.66) | 3.86 (0.68)
  id2, month 1: number analyzed (Participants) | 43 | 48
  id2, month 1 | 3.86 (0.70) | 3.83 (0.80)
  id2, month 3: number analyzed (Participants) | 38 | 44
  id2, month 3 | 3.77 (0.76) | 3.95 (0.77)
  id2, month 6: number analyzed (Participants) | 34 | 42
  id2, month 6 | 3.63 (0.84) | 3.87 (0.70)
  id2, month 9: number analyzed (Participants) | 29 | 37
  id2, month 9 | 3.83 (0.69) | 3.96 (0.61)
  id2, month 12: number analyzed (Participants) | 28 | 32
  id2, month 12 | 3.71 (0.73) | 3.91 (0.52)
Statistical Analysis 1: Comparison: Standard Foot Care Education vs Enhanced Foot Care Education; Test type: Equivalence — This trial aims to show the new treatment is no better and no worse; p = 0.6638, Mixed Models Analysis — The threshold of significance level set at 0.05

3. Secondary Outcome: Foot Complications
Description: Number of participants with foot complications
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Foot Care Education | Enhanced Foot Care Education
Number analyzed (Participants) | 48 | 51
Participants
  pre-ulcerative lesions | 7 | 11
  foot ulcer | 3 | 3
  subungual hematoma | 13 | 6
Statistical Analysis 1: Comparison: Standard Foot Care Education vs Enhanced Foot Care Education; Test type: Equivalence — The test will compare the number of complications between the two groups; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Standard Foot Care Education | Enhanced Foot Care Education
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/51
Other Adverse Events (participants affected / at risk) | 21/48 | 30/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Foot Care Education (N=48) | Enhanced Foot Care Education (N=51)
cellulitis, foot (Infections and infestations) | 0 (0) | 0 (0)
lower limb amputation (Infections and infestations) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Foot Care Education (N=48) | Enhanced Foot Care Education (N=51)
diabetic foot ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) — Diabetic foot ulcer, clean and not infected
Pre-ulcerative lesion (Skin and subcutaneous tissue disorders) | 7 (7) | 11 (11)
Ingrown (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Hospitalization (Cardiac disorders) | 8 (8) | 12 (12) — Nonstudy related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes